CLINICAL TRIAL: NCT06773312
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Efficacy and Pharmacokinetics of BC001 in Combination with Sintilimab and XELOX in the Treatment of HER-2 Negative Advanced or Metastatic Gastric Cancer or Gastroesophageal Junction Adenocarcinoma (GC/GEJ).
Brief Title: BC001 in Combination with Sintilimab and XELOX in the Treatment of HER-2 Negative Advanced or Metastatic Gastric Cancer or Gastroesophageal Junction Adenocarcinoma.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Luzhou Buchang Biopharmaceutical Co., Ltd. (Industry)
Collaborators: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BC001-GC/GEJ-102
Record Dates: First submitted 2025-01-02; First posted 2025-01-14 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Advanced or Metastatic Gastric Cancer; Gastroesophageal Junction Adenocarcinoma
Keywords: gastroesophageal junction adenocarcinoma; VEGFR2; gastric cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BC001+Sintilimab+XELOX (Experimental): BC001+Sintilimab+XELOX
  Interventions: Biological: BC001+Sintilimab+XELOX

INTERVENTIONS:
Biological: BC001+Sintilimab+XELOX — patients will be given : BC001 8mg/kg, 12mg/kg or 16mg/kg intravenously once every three weeks; Sintilimab 3mg/kg（body weight<60kg）or 200mg（body weight≥60kg）intravenously once every three weeks; Oxaliplatin 130mg/m2 intravenously once every three weeks; Capecitabine 1000mg/m2 orally once daily in the first two weeks of each three-week treatment cycle.

SUMMARY:
The goal of this clinical trial is to learn the efficaty and safety of BC001 in combination with Sintilimab and XELOX in treating patients with advanced or metastatic GC/GEJ.

Participants will:

Be administered with BC001, Sintilimab and Oxaliplatin once every three weeks for up to 24 months or until disease progression as per RECIST 1.1 or withdrawal from this study.

Take Capecitabine once daily in the first two weeks of each three-week treatment cycle for up to 24 months or until disease progression as per RECIST 1.1 or withdrawal from this study.

DETAILED DESCRIPTION:
This trial is an open-label Phase I clinical trial, which is divided into the dose escalation phase and the dose expansion phase. It aims to evaluate the safety, tolerability, pharmacokinetic (PK) characteristics and preliminary efficacy of BC001 in combination with Sintilimab and XELOX, and to determine the recommended Phase 2 dose (RP2D) and preliminary efficacy of BC001 in combination with Sintilimab and XELOX in the treatment of patients with HER-2 negative advanced or metastatic gastric cancer or gastroesophageal junction adenocarcinoma (GC/GEJ) who have never received systemic treatment before.

The dose escalation phase adopts a 3+3 dose escalation design and three dose groups are planned initially.

The dose expansion study will recommend two appropriate dose groups based on data from the dose escalation phase, and 30 subjects planned to be enrolled in each group. According to the safety and efficacy of each group, one of the doses will be selected and determined as the recommended Phase 2 dose (RP2D).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be able to understand and voluntarily sign the written informed consent.
2. Subjects must be willing and able to complete the study procedures and follow-up examinations.
3. Male or female subjects aged between 18 and 75 years old (including 18 and 75 years old).
4. HER-2 negative patients with advanced or metastatic gastric cancer or gastroesophageal junction adenocarcinoma (GC/GEJ) (according to the 8th edition of AJCC/UICC TNM staging) confirmed by histopathology or cytopathology, who have never received systemic treatment before (the time interval from the end of previous neoadjuvant treatment/adjuvant treatment to the recurrence of the disease > 6 months will be regarded as untreated).
5. According to RECIST version 1.1, there must be at least one measurable tumor lesion shown by CT or MRI examination.
6. Subjects with normal oral intake.
7. ECOG (Eastern Cooperative Oncology Group) performance score of 0 - 1.
8. Expected survival period is greater than 3 months.
9. There is no serious hematological, hepatic or renal function abnormality, meeting the following laboratory test results: the absolute neutrophil count (ANC) should be ≥1.5×10⁹/L, platelet (PLT) ≥100×10⁹/L, and hemoglobin (HGB) ≥90g/L; Serum creatinine (Cr) ≤1.5× the upper limit of normal range (ULN). When Cr > 1.5×ULN, , and creatinine clearance rate (Ccr)≥ 60mL/min(calculated according to the Cockcroft - Gault formula); the qualitative urine protein should be ≤1 +, or if the qualitative urine protein ≥2 +, the 24-hour urine protein < 1g; total bilirubin (TBIL) ≤1.5×ULN or ≤3×ULN (for patients with liver cancer or liver metastases), alanine aminotransferase (AST) and aspartate aminotransferase (ALT) ≤3.0×ULN or ≤5×ULN (for patients with liver cancer or liver metastases), alkaline phosphatase (ALP) ≤2.5×ULN or ≤5×ULN (for patients with liver cancer or liver metastases); the international normalized ratio (INR) or prothrombin time T (PT) ≤1.5×ULN, and the activated partial thromboplastin time (APTT) ≤1.5×ULN.
10. Male or female subjects should take effective contraceptive measures during the treatment period and within 6 months after the last dose administration.

Exclusion Criteria:

1. Subjects who have undergone major organ surgical operations (excluding needle biopsy) or had significant trauma within 4 weeks prior to the first use of the study drug, or who need to undergo elective surgeries during the trial period.
2. Subjects whose original lesions have invaded the central nervous system (CNS) with symptoms, are unstable or require high-dose steroids (≥10mg dexamethasone or equivalent dose) to achieve control.
3. Subjects suffering from other primary malignancies, except for malignancies with low metastasis risk and low death risk (5-year survival rate > 90%), such as malignancies that have been cured and have not relapsed within 3 years before enrollment in the study; completely resected basal cell and squamous cell skin cancers; completely resected carcinomas in situ of any type.
4. Subjects with active infections (such as viral, bacterial or fungal infections) that require systemic treatment.
5. Subjects currently suffering from interstitial lung disease (except for radiation-induced pulmonary fibrosis that does not require hormone treatment).
6. Subjects with a history of active bleeding within the past 4 weeks or at risk of gastrointestinal perforation, or with a history of recent surgeries that have not healed or with a history of wound complications caused by surgical operations.
7. Subjects who had gastrointestinal bleeding within 3 months prior to the use of the study drug and without evidence verified by endoscopy or colonoscopy that they have recovered; subjects with severe gastrointestinal diseases within 2 weeks prior to the use of the study drug.
8. Subjects with a history of severe cardiovascular and cerebrovascular diseases, including but not limited to: Having severe cardiac rhythm or conduction abnormalities, such as ventricular arrhythmias requiring clinical intervention, grade II - III atrioventricular block, etc.; Having suffered from acute coronary syndrome, congestive heart failure, aortic dissection, stroke/TIA or other grade 3 or above cardiovascular and cerebrovascular events within 6 months prior to the first dose administration; Having heart failure of New York Heart Association (NYHA) class > II or left ventricular ejection fraction (LVEF) < 50%; Having a baseline QTcF interval corrected for heart rate calculated by the Fridericia formula > 450 msec (for males) and > 470 msec (for females); Having any factors that increase the risk of QTc prolongation or arrhythmia, such as heart failure, hypokalemia, congenital long QT syndrome, a family history of long QT syndrome or using any concomitant drugs known to prolong the QT interval.

   Having a diastolic blood pressure ≥ 100 mmHg or a systolic blood pressure ≥ 160 mmHg after standardized treatment.
9. Subjects who have received treatments such as colony-stimulating factors and erythropoietin within 2 weeks prior to the use of the study drug.
10. Subjects who have been vaccinated with live vaccines within 4 weeks prior to the use of the study drug. Live vaccines include but are not limited to the following: measles, mumps, rubella, varicella/zoster (chickenpox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG) and typhoid vaccines. Seasonal influenza vaccines for injection are usually inactivated virus vaccines, so their use is permitted; intranasal influenza vaccines (e.g., FluMist) are attenuated live vaccines and are not permitted for use.
11. Subjects who are currently receiving long-term treatment with non-steroidal anti-inflammatory drugs (such as indomethacin, ibuprofen, etc.) or antiplatelet drugs (such as clopidogrel, ticlopidine, dipyridamole, etc.) (the use of aspirin is permitted with a maximum daily dose of 325mg).
12. Subjects with a known history of liver diseases of significant clinical significance, including active hepatitis (hepatitis B surface antigen positive and the copy number of HBV DNA > the normal value of the testing unit; hepatitis C virus antibody positive and the copy number of HCV RNA > the normal value of the testing unit), hepatic encephalopathy, hepatorenal syndrome, liver function at Child-Pugh grade B or more severe cirrhosis.
13. Subjects with a history of human immunodeficiency virus infection or suffering from other acquired or congenital immunodeficiency diseases.
14. Subjects who are preparing for or have previously received tissue/organ transplantation.
15. Subjects known to be allergic to the study drugs, monoclonal antibodies and other therapeutic protein preparations (fresh or frozen plasma, human serum albumin, cytokines, interleukins, etc.).
16. Subjects known to have alcohol and/or drug dependence.
17. Female subjects with a positive blood pregnancy test or those who are breastfeeding.
18. Subjects with known signs of active bleeding in the lesions.
19. Subjects with pleural effusion, pericardial effusion or ascites that are uncontrollable and require repeated drainage or medical intervention. Only those with a small amount of ascites shown by imaging but without symptoms can be enrolled.
20. Subjects known to have dihydropyrimidine dehydrogenase (DPD) deficiency (or those who have experienced grade 3 or above mucosal toxicity during previous fluorouracil-containing treatments).
21. Subjects with cardiac obstruction, pyloric obstruction or persistent and repeated vomiting (defined as vomiting ≥ 3 times within 24 hours).
22. Subjects who had intestinal obstruction or the following diseases within 3 months prior to the first use of the study drug: inflammatory bowel disease or extensive bowel resection (partial colectomy or extensive small bowel resection accompanied by chronic diarrhea), Crohn's disease, ulcerative colitis.
23. Subjects with a history of deep vein thrombosis, pulmonary embolism or any other serious thromboembolism within 3 months before enrollment; subjects who need to use vitamin K antagonists for anticoagulation or need to use heparin at a therapeutic dose (prophylactic dose is acceptable) during the study period.
24. Subjects who need to use systemic immunosuppressive therapy within 14 days prior to the first use of the study drug or during the study period, except for the following situations: intranasal, inhaled, topical steroids or local steroid injections (such as intra-articular injection); physiological doses of systemic corticosteroids (≤10mg/day prednisone or equivalent dose); short-term (≤7 days) use of steroids for the prevention or treatment of non-autoimmune allergic diseases.
25. Subjects judged by the researcher as being unsuitable for participating in this study for other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Adverse events | Through study completion, assessed up to 2 years
  The frequency, severity of adverse events during the trial.
Maximum tolerated dose（dose escalation phase） | Until the completion of the DLT (dose-limiting toxicity) observation period, about 21 days.
Recommended Phase 2 Dose(expansion phase) | Through study completion, assessed up to 2 years

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | 3 months
VEGF concentration in serum | 3 months
Immunogenicity | 3 months
  Anti-BC001 antibody.
Objective response rate (ORR) | Up to 2 years
  Defined as the proportion of patients who have a complete response (CR) or a partial response (PR) per RECIST 1.1.
Area under the curve (AUC) | 3 months
sVEGFR in serum | 3 months
sPD-L1 in serum | 3 months
Progression-free survival （PFS） | Up to 2 years
  The time interval from the start of the first drug administration to progressive disease per RECIST 1.1 or death from any cause
Overall survival (OS) | Up to 5 years
  The time interval from the first drug administration to death due to any cause.
Duration of response (DoR) | Up to 2 years
  The time interval from the first discovery of disease remission (CR or PR) to progressive disease per RECIST 1.1 or death from any cause
Disease control rate (DCR) | Up to 2 years
  Defined as the proportion of subjects who achieved a best response of Complete Response (CR), Partial Response (PR), or Stable Disease (SD) per RECIST 1.1.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No